CLINICAL TRIAL: NCT03446040
Title: A Phase 1/2 First-in-Human Study of BMS-986258 Alone and in Combination With Nivolumab in Advanced Malignant Tumors
Brief Title: An Investigational Immunotherapy Study of BMS-986258 Alone and in Combination With Nivolumab in Participants With Solid Cancers That Are Advanced or Have Spread
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA031-002; 2019-000442-35 (EudraCT Number)
Record Dates: First submitted 2018-02-21; First posted 2018-02-26 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A Dose Escalation: BMS-986258 (Experimental)
  Interventions: Biological: BMS-986258
- Part A1: BMS-986258 + Recombinant human hyaluronidase PH20 (rHuPH20) (Experimental)
  Interventions: Biological: BMS-986258; Drug: rHuPH20
- Part B Dose Escalation: BMS-986258 + nivolumab (Experimental)
  Interventions: Biological: BMS-986258; Biological: Nivolumab
- Part C Cohort Expansion: BMS-986258 + nivolumab (Experimental)
  Interventions: Biological: BMS-986258; Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986258 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part B Dose Escalation: BMS-986258 + nivolumab; Part C Cohort Expansion: BMS-986258 + nivolumab
Drug: rHuPH20 — Specified dose on specified days
  Other Names: Enhanze
  Arms: Part A1: BMS-986258 + Recombinant human hyaluronidase PH20 (rHuPH20)

SUMMARY:
The purpose of this study is to determine whether BMS-986258 both monotherapy and in combination with Nivolumab is safe and tolerable in the treatment of advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of one of the 5 tumors [renal cell carcinoma (RCC), colorectal cancer (CRC), non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), triple negative breast cancer (TNBC)] (metastatic, recurrent, and/or unresectable), with measurable disease per response evaluation criteria in solid tumors v1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Participants must have received, and then progressed, relapsed, or been intolerant to, at least 1 standard treatment regimen in the advanced or metastatic setting according to solid tumor histologies
* Women must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Active, known or suspected autoimmune disease
* Cytotoxic agents, unless at least 4 weeks have elapsed from last dose of prior anti-cancer therapy and initiation of study therapy
* Other active malignancy requiring concurrent intervention

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (10):
  - Local Institution - 0004, Los Angeles, California
  - Local Institution - 0006, Los Angeles, California
  - Local Institution - 0007, Aurora, Colorado
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Local Institution - 0018, Ann Arbor, Michigan
  - Local Institution - 0010, Grand Rapids, Michigan
  - Local Institution - 0012, Lebanon, New Hampshire
  - Local Institution - 0016, Cincinnati, Ohio
  - Local Institution - 0005, Pittsburgh, Pennsylvania
  - Local Institution - 0002, Germantown, Tennessee
- Australia (2):
  - Local Institution - 0013, Westmead, New South Wales
  - Local Institution - 0015, Melbourne, Victoria
- Canada (2):
  - Local Institution - 0014, Edmonton, Alberta
  - Local Institution - 0019, Vancouver, British Columbia
- Japan (2):
  - Local Institution - 0009, Kobe, Hyōgo
  - Local Institution - 0008, Chuo-ku, Tokyo

REFERENCES:
- [Derived] El Halabi L, Adam J, Gravelle P, Marty V, Danu A, Lazarovici J, Ribrag V, Bosq J, Camara-Clayette V, Laurent C, Ghez D. Expression of the Immune Checkpoint Regulators LAG-3 and TIM-3 in Classical Hodgkin Lymphoma. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):257-266.e3. doi: 10.1016/j.clml.2020.11.009. Epub 2020 Nov 12. PMID 33277223
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were treated in Part A, Part A1, and Part B. No participants were enrolled or treated in Part C. 4 participants in Part A1 transitioned to Part B.
Groups:
- Part A: BMS-986258 8 mg: Participants received 8 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 24 mg: Participants received 24 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 72 mg: Participants received 72 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 200 mg: Participants received 200 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 480 mg: Participants received 480 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 800 mg: Participants received 800 mg BMS-986258 IV every 4 weeks (Q4W) for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 1200 mg: Participants received 1200 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 1600 mg: Participants received 1600 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A: BMS-986258 2400 mg: Participants received 2400 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part B: BMS-986258 480 mg + NIVO 480 mg: Participants received 480 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part B: BMS-986258 800 mg + NIVO 480 mg: Participants received 800 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part B: BMS-986258 1200 mg + NIVO 480 mg: Participants received 1200 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part B: BMS-986258 1600 mg + NIVO 480 mg: Participants received 1600 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A1: BMS-986258 1200 mg + ENHANZE: Participants received 1200 mg BMS-986258 with rHuPH20 (ENHANZE) SC for the first dose in Cycle 1. All subsequent doses of BMS-986258 were received as monotherapy IV, every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
Period: Overall Study
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Started (Started = Treated) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 11 | 4 | 15 | 15
Transitioned From Part A1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 8 | 6
Not Completed | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 4 | 4 | 10 | 4 | 7 | 9
Not completed — Disease progression | 3 | 3 | 3 | 4 | 4 | 6 | 3 | 4 | 2 | 4 | 9 | 3 | 7 | 7
Not completed — Study drug toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Participant requested to discontinue study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 11 | 4 | 15 | 15 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (16.17) | 45.7 (6.03) | 61.5 (3.11) | 67.0 (4.24) | 60 (12.44) | 61.1 (7.10) | 65.3 (8.33) | 54.8 (8.07) | 58.4 (5.85) | 64.5 (5.07) | 62.5 (7.75) | 57.3 (16.2) | 58.5 (15.0) | 57.8 (12.27) | 59.6 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 3 | 1 | 4 | 3 | 1 | 2 | 2 | 3 | 2 | 5 | 4 | 35
  Male | 2 | 3 | 0 | 1 | 3 | 5 | 0 | 4 | 6 | 2 | 8 | 2 | 10 | 11 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 2 | 3 | 4 | 4 | 3 | 8 | 3 | 5 | 8 | 3 | 10 | 4 | 11 | 14 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 2 | 2 | 4 | 3 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 9
  White | 2 | 0 | 2 | 2 | 2 | 7 | 2 | 2 | 5 | 3 | 8 | 2 | 8 | 10 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any new untoward medical occurrence or worsening of a preexisting medical condition in a study participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
  A Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event)
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect.
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 78 weeks)
Population: All treated participants. Participants who started in the Part A1 group but transitioned to Part B are accounted for in both treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- Part A1: BMS-986258 1200 mg + ENHANZE: Participant received 1200 mg BMS-986258 with rHuPH20 (ENHANZE) SC for the first dose in Cycle 1. All subsequent doses of BMS-986258 were received as monotherapy IV, every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 11 | 6 | 17 | 15
Participants
  Adverse Events (AEs) | 3 | 3 | 4 | 4 | 4 | 8 | 2 | 5 | 8 | 4 | 11 | 6 | 17 | 13
  Serious Adverse Events (SAEs) | 1 | 2 | 3 | 1 | 0 | 4 | 1 | 3 | 2 | 2 | 6 | 1 | 6 | 3
  Adverse Events (AEs) leading to discontinuation of study treatment | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

2. Primary Outcome: Number of Participants Who Died During the Study
Description: The number of participants who died during the study.
Time Frame: From first dose until death due to any cause (up to approximately 78 months)
Population: All treated participants. Participants who crossed over from part A1 are accounted for under their original arm assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 11 | 4 | 15 | 15
Participants | 3 | 3 | 3 | 3 | 3 | 7 | 3 | 4 | 5 | 3 | 9 | 0 | 10 | 8

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose-limiting toxicity (DLT) refers to a side effect or adverse reaction caused by a drug that is severe enough to prevent an increase in dose or level of that drug. It is typically identified during clinical trials to determine the highest dose of a drug that can be given safely without causing unacceptable side effects.
  A participant was considered DLT evaluable if they received 1 dose of BMS-986258 in Part A or 1 dose of BMS-986258 and nivolumab 480mg in Part B and completed the DLT observation period.
  Participants who withdraw from the study during the 4-week DLT evaluation period for reasons other than a DLT may be replaced with a new participant at the same dose level.
Time Frame: From first dose (Cycle 1 Day 1) until day 28 (Cycle 1 Day 28)
Population: All treated participants who were evaluable for DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 5 | 3 | 5 | 2 | 5 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percent of treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) per RECIST v1.1.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose until disease progression or death, whichever occurred first (up to approximately 78 months)
Population: All treated participants. Prespecified to be reported collectively per Part. Participants who crossed over from part A1 to Part B are accounted for in both arms.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Part A: All Doses: Participants received BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks))
- Part B: All Doses: Participants received BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks))
Arm/Group | Part A: All Doses | Part B: All Doses | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 43 | 37 | 15
Percent of Participants | 0 [0.00 to 8.22] | 5.4 [0.66 to 18.19] | 0 [0.00 to 21.80]

5. Secondary Outcome: Median Duration of Response (mDOR)
Description: Median duration of response (mDOR) for a participant with a best overall response (BOR) of complete response (CR) or partial response (PR) is defined as the time between the date of first response and the date of the first objectively documented disease progression (DP) per RECIST v1.1 or death, whichever occurred first.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Disease Progression (DP): At least a 20% increase in the sum of the diameters of target lesions, with an absolute increase of at least 5 mm, or the appearance of new lesions.
  Based on Kaplan-Meier estimates.
Time Frame: From first dose until disease progression or death whichever occurred first (up to approximately 78 months)
Population: All treated participants witha complete or partial response. Prespecified to be reported collectively per Part. Response evaluable participants who crossed over from part A1 to Part B are accounted for in both arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: All Doses | Part B: All Doses | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 0 | 2 | 0
Months |  | NA [NA to NA] — Insufficient number of events to calculate median, LL, and UL by K-M methodology. |

6. Secondary Outcome: Progression-Free Survival (PFS) Rate at 6, 9, and 12 Months
Description: Progression free survival (PFS) for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurred first.
  Disease Progression (DP): At least a 20% increase in the sum of the diameters of target lesions, with an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: At 6, 9, and 12 months after first dose
Population: All treated participants. Prespecified to be reported collectively per Part. Treated participants who crossed over from part A1 to Part B are accounted for in both arms.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Part A: All Doses | Part B: All Doses | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 43 | 37 | 15
Percent of Participants
  6-month | 21.4 [9.3 to 36.8] | 21.9 [8.4 to 39.3] | 8.7 [0.5 to 32.0]
  9-month | 17.1 [6.2 to 32.6] | 8.2 [0.8 to 27.7] | 8.7 [0.5 to 32.0]
  12-month | 17.1 [6.2 to 32.6] | 0.0 [NA to NA] — 95% CI not calculated as PFS-Rate = 0% | 0.0 [NA to NA] — 95% CI not calculated as PFS-Rate = 0%

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of BMS-986258
Description: Cmax (Maximum Concentration) is the highest level of a drug in the blood after it has been taken. It shows the peak level of the drug, which helps in understanding how much of the drug is absorbed and how strong its effects might be.
Time Frame: Part A and B: On Cycle 1 Day 1 and Cycle 3 Day 1 (1 cycle = 8 weeks); Part A1: On Cycle 1 Day 1 and Cycle 1 Day 29 (1 cycle = 8 weeks)
Population: All treated participants with available PK results. PK evaluable participants who crossed over from Part A1 to Part B are accounted for in both arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 10 | 3 | 15 | 9
ug/mL
  Cycle 1 Day 1 | 2.27 (53.8) | 5.34 (36.2) | 31.5 (10.9) | 47.2 (120) | 121 (30.7) | 239 (35.6) | 423 (12.9) | 412 (26.7) | 890 (29.2) | 154 (43.4) | 244 (24.8) | 449 (31.5) | 579 (19.4) | 121 (44.1)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 2 | 7 | 0
  Cycle 3 Day 1 |  | 9.26 (NA) — Insufficient number of participants to calculate geometric CV |  | 50 (NA) — Insufficient number of participants to calculate geometric CV |  | 356 (NA) — Insufficient number of participants to calculate geometric CV |  |  | 605 (NA) — Insufficient number of participants to calculate geometric CV | 111 (NA) — Insufficient number of participants to calculate geometric CV | 161 (NA) — Insufficient number of participants to calculate geometric CV | 422 (NA) — Insufficient number of participants to calculate geometric CV | 684 (18.1) |
  Cycle 1 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  | 479 (21.2)

8. Secondary Outcome: Area Under the Curve From Time 0 to T (AUC(0-T)) of BMS-986258
Description: AUC (0-T) is the total exposure to the drug over a specific period; from the time you take it until a specified time.
  It helps in understanding the overall amount of drug that has been in your body over that time period.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 10 | 3 | 15 | 9
h*ug/mL
  Cycle 1 Day 1 | 53.7 (50.8) | 457 (56) | 4690 (43.3) | 8180 (101) | 26100 (46.7) | 46000 (83.9) | 97000 (23.3) | 75300 (44.5) | 179000 (24.3) | 29000 (51.4) | 44300 (34.9) | 84100 (83.2) | 118000 (25.4) | 48500 (51.1)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 2 | 7 | 0
  Cycle 3 Day 1 |  | 1400 (NA) — Insufficient number of participants to calculate geometric CV |  | 13400 (NA) — Insufficient number of participants to calculate geometric CV |  | 102000 (NA) — Insufficient number of participants to calculate geometric CV |  |  | 135000 (NA) — Insufficient number of participants to calculate geometric CV | 29800 (NA) — Insufficient number of participants to calculate geometric CV | 38200 (NA) — Insufficient number of participants to calculate geometric CV | 89000 (NA) — Insufficient number of participants to calculate geometric CV | 171000 (27) |
  Cycle 1 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  | 138000 (21)

9. Secondary Outcome: Area Under the Curve Over the Dosing Interval AUC(TAU) of BMS-986258
Description: AUC(TAU) (Area Under the Curve over the Dosing Interval) is the total exposure to the drug over one complete dosing interval (the time between doses). It helps in understanding how much of the drug is in your body over the entire period between doses, which is important for determining the right dosing schedule.
Time Frame: Part A and B: 0 to 28 days post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (1 cycle = 8 weeks); Part A1: 0 to 28 days post-dose on Cycle 1 Day 1 and Cycle 1 Day 29 (1 cycle = 8 weeks)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 0 | 3 | 4 | 4 | 4 | 8 | 3 | 5 | 8 | 4 | 10 | 3 | 15 | 7
h*ug/mL
  Cycle 1 Day 1 |  | 587 (41.9) | 4870 (43.7) | 8400 (105) | 26900 (47.4) | 56400 (45) | 100000 (18) | 85800 (21.9) | 187000 (29.5) | 29000 (51.4) | 47300 (29.4) | 89600 (67.9) | 120000 (22.5) | 46200 (53.9)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 7 | 0
  Cycle 3 Day 1 |  | 1440 (NA) — Insufficient number of participants to calculate geometric CV |  | 13400 (NA) — Insufficient number of participants to calculate geometric CV |  | 102000 (NA) — Insufficient number of participants to calculate geometric CV |  |  | 135000 (NA) — Insufficient number of participants to calculate geometric CV | 18600 (NA) — Insufficient number of participants to calculate geometric CV | 38200 (NA) — Insufficient number of participants to calculate geometric CV | 89000 (NA) — Insufficient number of participants to calculate geometric CV | 172000 (26.1) |
  Cycle 1 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  | 134000 (17.3)

10. Secondary Outcome: Concentration at the End of the Dosing Interval (Ctau) of BMS-986258
Description: Ctau (Concentration at the End of the Dosing Interval) is the level of the drug in the blood just before the next dose is due. It shows how much of the drug remains in your body before taking the next dose, which helps in ensuring that the drug levels stay effective without dropping too low.
Time Frame: Part A and B: On Cycle 1 Day 29 and Cycle 3 Day 29 (1 cycle = 8 weeks); Part A1: On Cycle 1 Day 29 and Cycle 2 Day 1 predose (1 cycle = 8 weeks)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 0 | 3 | 4 | 4 | 4 | 8 | 3 | 5 | 8 | 4 | 10 | 3 | 15 | 7
ug/mL
  Cycle 1 Day 29 predose |  | 0.0245 (52.3) | 1.58 (116) | 2.59 (369) | 15.5 (68.6) | 37.2 (62.9) | 55.7 (55.2) | 36.9 (68.5) | 109 (44.6) | 15.6 (82.3) | 23.5 (70.3) | 39.8 (229) | 68.4 (47.1) | 37.7 (80.2)
  Cycle 3 Day 29 predose: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 7 | 0
  Cycle 3 Day 29 predose |  | 0.0711 (NA) — Insufficient number of participants to calculate geometric CV |  | 8.32 (NA) — Insufficient number of participants to calculate geometric CV |  | 80.3 (NA) — Insufficient number of participants to calculate geometric CV |  |  | 71.3 (NA) — Insufficient number of participants to calculate geometric CV | 7.77 (NA) — Insufficient number of participants to calculate geometric CV | 25 (NA) — Insufficient number of participants to calculate geometric CV | 37.1 (NA) — Insufficient number of participants to calculate geometric CV | 121 (36.6) |
  Cycle 2 Day 1 predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Cycle 2 Day 1 predose |  |  |  |  |  |  |  |  |  |  |  |  |  | 114 (13)

11. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of BMS-986258
Description: Tmax (Time to Reach Maximum Concentration) is the time it takes for the drug to reach its highest level in the blood after taking it. It helps in understanding how quickly the drug starts to work and reaches its peak effect.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 9 | 3 | 5 | 8 | 4 | 10 | 3 | 15 | 9
Hours
  Cycle 1 Day 1 | 0.808 [0.033 to 4] | 1.23 [0.117 to 4] | 1.4 [0.45 to 4] | 2.11 [0.45 to 24.5] | 3.92 [0.617 to 24] | 0.998 [0.467 to 4.13] | 1.09 [0.467 to 4.38] | 1.47 [1.47 to 1.48] | 3.11 [2 to 4.05] | 0.812 [0.467 to 4] | 4.18 [4 to 4.58] | 1.02 [0.983 to 1.07] | 2.29 [1.47 to 5.52] | 123 [72.2 to 168]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 2 | 7 | 0
  Cycle 3 Day 1 |  | 4 [4 to 4] |  | 0.7 [0.7 to 0.7] |  | 4.27 [4 to 4.55] |  |  | 2 [2 to 2] | 0.499 [0.467 to 0.533] | 0.467 [0.467 to 0.467] | 2.02 [1.02 to 4] | 2.74 [1.47 to 5.48] |
  Cycle 1 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.26 [0.967 to 2.33]

12. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to BMS-986258 or Nivolumab
Description: Baseline ADA-positive participant is defined as a participant who has an ADA-detected sample at baseline. ADA-positive participant is a participant with at least 1 ADA-positive sample relative to baseline after initiation of the treatment
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 78 weeks)
Population: All treated participants with baseline and at least one post-baseline pre-infusion ADA assessment. Prespecified to be reported collectively per Part. PK evaluable participants who crossed over from Part A1 to Part B are accounted for in both arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: All Doses | Part B: All Doses | Part A1: BMS-986258 1200 mg + ENHANZE
Number analyzed (Participants) | 35 | 28 | 14
Participants
  Baseline ADA positive: BMS-986258: number analyzed (Participants) | 35 | 27 | 14
  Baseline ADA positive: BMS-986258 | 0 | 0 | 0
  ADA positive: BMS-986258: number analyzed (Participants) | 35 | 27 | 14
  ADA positive: BMS-986258 | 2 | 0 | 0
  Baseline ADA positive: nivolumab: number analyzed (Participants) | 0 | 28 | 1
  Baseline ADA positive: nivolumab |  | 1 | 0
  ADA positive: nivolumab: number analyzed (Participants) | 0 | 28 | 1
  ADA positive: nivolumab |  | 2 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM) was assessed from first dose until death due to any cause (up to approximately 78 months). Serious-adverse events (AEs) and Other adverse events (AEs) were assessed from first dose until 100 days after last dose of study therapy (up to approximately 78 weeks).
Description: ACM, SAEs and AEs represent all treated participants. Prespecified for Part A1 crossover participants to be shown separately from those who did not crossover.
Groups:
- Part A: BMS-986258 8 mg: Participants received 8 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 24 mg: Participants received 24 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 72 mg: Participants received 72 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 200 mg: Participants received 200 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 480 mg: Participants received 480 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 800 mg: Participants received 800 mg BMS-986258 IV every 4 weeks (Q4W) for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 1200 mg: Participants received 1200 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 1600 mg: Participants received 1600 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A: BMS-986258 2400 mg: Participants received 2400 mg BMS-986258 IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part B: BMS-986258 480 mg + NIVO 480 mg: Participants received 480 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part B: BMS-986258 800 mg + NIVO 480 mg: Participants received 800 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part B: BMS-986258 1200 mg + NIVO 480 mg: Participants received 1200 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part B: BMS-986258 1600 mg + NIVO 480 mg: Participants received 1600 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A1: BMS-986258 1200 mg + ENHANZE: Participants received 1200 mg BMS-986258 with rHuPH20 (ENHANZE) SC for the first dose in Cycle 1. All subsequent doses of BMS-986258 were received as monotherapy IV, every 4 weeks (Q4W) twice per cycle for up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
- Part A1 Crossover to Part B: 1200 mg BMS + 480 mg Nivo: Participants received 1200 mg BMS-986258 with rHuPH20 (ENHANZE) SC for the first dose in Cycle 1. All subsequent doses of BMS-986258 were received as monotherapy IV, every 4 weeks (Q4W) twice per cycle. Upon crossover, participants received 1200 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for a total treatment duration of up to 96 weeks (12 treatment cycles (each cycle = 8 weeks)).
- Part A1 Crossover to Part B: 1600 mg BMS + 480 mg Nivo: Participants received 1200 mg BMS-986258 with rHuPH20 (ENHANZE) SC for the first dose in Cycle 1. All subsequent doses of BMS-986258 were received as monotherapy IV, every 4 weeks (Q4W) twice per cycle. Upon crossover, participants received 1600 mg BMS-986258 and 480 mg nivolumab IV every 4 weeks (Q4W) twice per cycle for a total treatment duration of up to 96 weeks (12 treatment cycles (each cycle = 8 weeks).
Arm/Group | Part A: BMS-986258 8 mg | Part A: BMS-986258 24 mg | Part A: BMS-986258 72 mg | Part A: BMS-986258 200 mg | Part A: BMS-986258 480 mg | Part A: BMS-986258 800 mg | Part A: BMS-986258 1200 mg | Part A: BMS-986258 1600 mg | Part A: BMS-986258 2400 mg | Part B: BMS-986258 480 mg + NIVO 480 mg | Part B: BMS-986258 800 mg + NIVO 480 mg | Part B: BMS-986258 1200 mg + NIVO 480 mg | Part B: BMS-986258 1600 mg + NIVO 480 mg | Part A1: BMS-986258 1200 mg + ENHANZE | Part A1 Crossover to Part B: 1200 mg BMS + 480 mg Nivo | Part A1 Crossover to Part B: 1600 mg BMS + 480 mg Nivo
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/4 | 3/4 | 3/4 | 7/9 | 3/3 | 4/5 | 5/8 | 3/4 | 9/11 | 0/4 | 10/15 | 7/11 | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/4 | 1/4 | 0/4 | 4/9 | 1/3 | 3/5 | 2/8 | 2/4 | 6/11 | 1/4 | 6/15 | 3/11 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 4/4 | 4/4 | 4/4 | 8/9 | 2/3 | 5/5 | 8/8 | 4/4 | 9/11 | 4/4 | 15/15 | 9/11 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BMS-986258 8 mg (N=3) | Part A: BMS-986258 24 mg (N=3) | Part A: BMS-986258 72 mg (N=4) | Part A: BMS-986258 200 mg (N=4) | Part A: BMS-986258 480 mg (N=4) | Part A: BMS-986258 800 mg (N=9) | Part A: BMS-986258 1200 mg (N=3) | Part A: BMS-986258 1600 mg (N=5) | Part A: BMS-986258 2400 mg (N=8) | Part B: BMS-986258 480 mg + NIVO 480 mg (N=4) | Part B: BMS-986258 800 mg + NIVO 480 mg (N=11) | Part B: BMS-986258 1200 mg + NIVO 480 mg (N=4) | Part B: BMS-986258 1600 mg + NIVO 480 mg (N=15) | Part A1: BMS-986258 1200 mg + ENHANZE (N=11) | Part A1 Crossover to Part B: 1200 mg BMS + 480 mg Nivo (N=2) | Part A1 Crossover to Part B: 1600 mg BMS + 480 mg Nivo (N=2)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asterixis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BMS-986258 8 mg (N=3) | Part A: BMS-986258 24 mg (N=3) | Part A: BMS-986258 72 mg (N=4) | Part A: BMS-986258 200 mg (N=4) | Part A: BMS-986258 480 mg (N=4) | Part A: BMS-986258 800 mg (N=9) | Part A: BMS-986258 1200 mg (N=3) | Part A: BMS-986258 1600 mg (N=5) | Part A: BMS-986258 2400 mg (N=8) | Part B: BMS-986258 480 mg + NIVO 480 mg (N=4) | Part B: BMS-986258 800 mg + NIVO 480 mg (N=11) | Part B: BMS-986258 1200 mg + NIVO 480 mg (N=4) | Part B: BMS-986258 1600 mg + NIVO 480 mg (N=15) | Part A1: BMS-986258 1200 mg + ENHANZE (N=11) | Part A1 Crossover to Part B: 1200 mg BMS + 480 mg Nivo (N=2) | Part A1 Crossover to Part B: 1600 mg BMS + 480 mg Nivo (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 3 | 0 | 3 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 4 | 1 | 2 | 1 | 2 | 2
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 1 | 2 | 4 | 1 | 1 | 3 | 1 | 6 | 0 | 4 | 3 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drain site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 2 | 5 | 0 | 3 | 1 | 2 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 4 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03446040/Prot_SAP_000.pdf